CLINICAL TRIAL: NCT06684626
Title: The Role of Butirprost® as an Adjuvant in Enhancing the Effect of Antibiotics in Patients Affected by Chronic Bacterial Prostatitis: A Randomized Prospective Trial
Brief Title: The Role of Butirprost® in Combination With Antibiotics in Chronic Bacterial Prostatitis (CBP) Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Benito Fabio Mirto, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 156.2023
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Prostate Inflammation; Prostate Disease; Chronic Bacterial Prostatitis
Keywords: BACTERIAL PROSTATITIS; ANTIBIOTICS; LUTS; QoL; IPSS; Hyaluronic acid
MeSH Terms: conditions — Prostatitis; Prostatic Diseases | interventions — Hyaluronic Acid; Levofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butirprost and antibiotic (Experimental): The treatment schedule was based on fluoroquinolone (levofloxacin, 1 tablet 500 mg daily for 4 weeks) plus 1 tablet of Butirprost® daily for 4 weeks
  Interventions: Drug: Sodium Hyaluronate; Drug: Levofloxacin 500mg
- Antibiotic (Active Comparator): the treatment schedule was based on oral fluoroquinolone only (levofloxacin, 1 tablet 500 mg daily for 4 weeks)
  Interventions: Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Sodium Hyaluronate — Sodium Hyaluronate (Butirprost®) is a nutraceutical formulation in suppository form, designed for the management of chronic bacterial prostatitis (CBP). It contains key ingredients such as sodium hyaluronate, a derivative of hyaluronic acid (HA), along with Plantago major. Sodium hyaluronate is valued for its potent anti-inflammatory and tissue-regenerative properties, while Plantago major offers additional benefits through its soothing and wound-healing effects, enhancing the overall efficacy of the formulation in treating CBP.
  Other Names: Butirprost®
  Arms: Butirprost and antibiotic
Drug: Levofloxacin 500mg — Treatment typically involves fluoroquinolones alone, such as levofloxacin.

SUMMARY:
Bacterial prostatitis (BP) is a common prostatic infection characterized by pain and urinary symptoms, often with negative bacterial cultures from prostatic secretions. It affects young and older men bimodally and significantly impacts quality of life (QoL). Treatment typically involves antibiotics, but a multimodal approach with additional nutraceuticals may enhance outcomes. This work aims to assess the efficacy of Butirprost® in association with fluoroquinolones in patients with Chronic Bacterial Prostatitis (CBP).

ELIGIBILITY:
Inclusion Criteria:

* patient aged between 18 and 50 years
* symptoms consistent with CBP
* positive Mears-Stamey test

Exclusion Criteria:

* patients younger than 18 years
* history of neurological disease, urinary stones or cancer
* allergy to fluoroquinolones or any components of Butirprost®
* post-void residual > 50 mL
* Use of alpha-blockers or 5-alpha-reductase inhibitors (5-ARI)
* previous prostatic surgery, antibiotic treatment within four weeks prior to the study
* refusal to provide informed consent and incomplete follow-up data
* Patients testing positive for certain pathogens like Chlamydia trachomatis (Ct), Ureaplasma urealyticum, Neisseria gon-orrhoeae, herpes simplex virus types 1 and 2 (HSV-1/2), and human papillomavirus (HPV)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in pain | 30 days
  Assessing the National Institute of Health-Chronic Prostatitis Symptom Index (0-31) and its pain subset at 15- and 30 days (lower scores mean better outcomes).
Change in urinary symptoms | 30 days
  Assessing the National Institute of Health-Chronic Prostatitis Symptom Index (0-31) and its urinary subset at 15- and 30 days (lower scores mean better outcomes).
Change in Quality of Life (QoL) | 30 days
  Assessing the National Institute of Health-Chronic Prostatitis Symptom Index (0-31) its subsets at 15- and 30 days (lower scores mean better outcomes).
Change in Quality of Life (QoL) | 30 days
  Assessing the International Prostatic Symptoms Score (0-35) and its subsets at 15- and 30 days (lower scores mean better outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Napoli, Italy